CLINICAL TRIAL: NCT05443243
Title: Is a THA Stem in Varus a Risk Factor of Long-term Mechanical Complication
Acronym: PTHVarus
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PTHVarus ( 29BRC22.0081)
Record Dates: First submitted 2022-05-17; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-04

CONDITIONS: Hip Arthritis
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Varus Stems: Patients with a THA Stem implanted in Varus position
  Interventions: Procedure: Total Hip Arthroplasty
- Neutral stems: Patients with a THA Stem implanted in Neutral position
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Patient were operated, a Total hip arthroplasty was performed

SUMMARY:
The objective of this study is to compare the long-term survival as well as the functional and radiographic results of the rods in the alignment of the varus to the stems in the neutral alignment by comparing 2 groups of implanted Total Hip Arthroplasty. 1 group of stems implanted in varus position. 1 group of stems implanted in neutral position

DETAILED DESCRIPTION:
ABSTRACT:

Introduction: Femoral stem positioning in the frontal plane has always been considered a fundamental criterion for implant survival and for functional and radiographic outcomes in total hip arthroplasty (THA). The impact of implanting cementless femoral stems in varus alignment on long-term mechanical complications remains poorly defined in the literature. The aim of our study is to compare long-term survivorship as well as functional and radiographic outcomes of stems in varus alignment to stems in neutral alignment.

Patients and Methods: This single center, multi-surgeon, retrospective case-control study will compare a group of 105 THA patients with varus stem alignment (VS) to a control group of 105 THA patients with neutral stem alignment (NS), operated in Brest center between January 2007 and December 2012. The primary outcome measure is implant survival. Secondary outcomes include functional outcomes: HHS, PMA, thigh pain, dislocation and hip ROM; and radiographic outcomes: radiolucency, Agora Roentgenography Assessment (ARA) score, osseointegration, heterotopic ossification, subsidence and stress shielding.

ELIGIBILITY:
Inclusion Criteria:

* PTH rod implanted in varus,
* Having X-rays and clinical data in their file
* Within a period of less than 6 months
* No opposition

Exclusion Criteria:

* PTH in a context of fracture of the femoral neck
* PTH 2nd intention
* Lost to sight
* Patients who died within 6 months
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a first-line PTH between 2007 and 2012,
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Survival rate | It was measured in October 2021
  The main outcome measured was the survival of the implant

SECONDARY OUTCOMES:
HHS | It was measured in October 2021
  Functional outcome : - The Harris Hip Score (HHS) [26] which assesses pain, function, deformity and range of motion (ROM) with a maximum score of 100
PMA score : | It was measured in October 2021
  Functional outcome : which assesses pain, gait and mobility with a maximum score of 18
Thigh pain | It was measured in October 2021
  Functional outcome : we measured the rate of patients experiencing pain at the level of the thigh
Dislocation | It was measured in October 2021
  Functional outcome : hip disclocation rate over the follow up period
Hip ROM | It was measured in October 2021
  Functional outcome : Hip range of motion in flexion, adduction, extension, abduction and rotations
Radiolucency | It was measured in October 2021
  Radiographic outcome : - Radiolucency according to the Gruen/Callaghan zones
Agora Roentgenography Assessment (ARA) score | It was measured in October 2021
  Radiographic outcome : - Agora Roentgenography Assessment (ARA) score for cementless femoral stem stability according to Epinette
Osseointegration | It was measured in October 2021
  Radiographic outcome mesured was described in "Roentgenographic assessment of the biologic fixation of porous-surfaced femoral components" Engh CA, Massin P, Suthers KE"
Heterotopic ossification | t was measured in October 2021
  Radiographic outcome : - Brooker classification of heterotopic ossification
Subsidence | t was measured in October 2021
  Radiographic outcome : - Subsidence: considered significant if more than 5 mm between the immediate postoperative x-ray and the last follow-up x-ray. Subsidence was assessed by measuring the distance between the tip of the trochanter and the "shoulder" of the stem
Stress shielding. | t was measured in October 2021
  Radiographic outcome : we measured the rate of patients with Xray showing stress shielding signs

CONTACTS AND LOCATIONS:
Overall Officials: Hoel Letissier, MD, Principal Investigator — CHU de Brest
Locations (1):
- CHU de Brest, Brest, France

REFERENCES:
- [Result] Batailler C, Fary C, Servien E, Lustig S. Influence of femoral broach shape on stem alignment using anterior approach for total hip arthroplasty: A radiologic comparative study of 3 different stems. PLoS One. 2018 Oct 5;13(10):e0204591. doi: 10.1371/journal.pone.0204591. eCollection 2018. PMID 30289882
- [Result] Murphy CG, Bonnin MP, Desbiolles AH, Carrillon Y, Asmall yi, Ukrainiant Si Selmi T. Varus will have varus; a radiological study to assess and predict varus stem placement in uncemented femoral stems. Hip Int. 2016 Nov 10;26(6):554-560. doi: 10.5301/hipint.5000412. Epub 2016 Oct 15. PMID 27768218
- [Result] Fottner A, Woiczinski M, Kistler M, Schroder C, Schmidutz TF, Jansson V, Schmidutz F. Varus malalignment of cementless hip stems provides sufficient primary stability but highly increases distal strain distribution. Clin Biomech (Bristol). 2018 Oct;58:14-20. doi: 10.1016/j.clinbiomech.2018.07.006. Epub 2018 Jul 5. PMID 30005422